CLINICAL TRIAL: NCT00036634
Title: A Phase 1/2, Randomized, Double-Blind, Active Controlled, Dose Escalation Study of the Safety, Tolerance, Pharmacokinetic,, and Antiviral Activity of GS-7340-02 in Antiretroviral-Naive Patients Who Are Chronically Infected With HIV-1
Brief Title: A Dose Escalation Study of Tenofovir Alafenamide in Treatment-Naive Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-120-1101
Record Dates: First submitted 2002-05-13; First posted 2002-05-14 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: HIV Infections
Keywords: treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Tenofovir DF (Active Comparator): Participants received tenofovir DF 300 mg for 14 days
  Interventions: Drug: Tenofovir DF
- Tenofovir alafenamide 50 mg (Experimental): Participants received tenofovir alafenamide 50 mg for 14 days
  Interventions: Drug: Tenofovir alafenamide
- Tenofovir alafenamide 150 mg (Experimental): Participants received tenofovir alafenamide 150 mg for 14 days
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Tenofovir DF — Tenofovir DF tablet administered orally once daily
  Other Names: Viread®
  Arms: Tenofovir DF
Drug: Tenofovir alafenamide — Tenofovir alafenamide tablet(s) administered orally once daily
  Other Names: GS-7340
  Arms: Tenofovir alafenamide 150 mg; Tenofovir alafenamide 50 mg

SUMMARY:
This study evaluated two doses of tenofovir alafenamide versus tenofovir disoproxil fumarate (tenofovir DF).

ELIGIBILITY:
Inclusion Criteria

* HIV-1 RNA levels greater than or equal to 30,000 copies/mL
* CD4 count greater than or equal to 200 cells/mm3
* Serum creatinine <1.5 mg/dl
* Hepatic transaminases less than or equal to 2.5 times the upper limit of normal
* Total bilirubin less than or equal to 1.5 mg/dL
* Adequate hematologic function
* Serum amylase less than or equal to 1.5 times the upper limit of normal
* Serum phosphate greater than or equal to 2.2 mg/dL
* Not pregnant

Exclusion Criteria

* Prior treatment with antiretroviral therapy
* Immunization within 30 days of study entry
* A new AIDS defining condition within 30 days of study entry
* Receiving nephrotoxic agents, probenecid, chemotherapeutic agents, corticosteroids, interleukin-2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-03; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Time-weighted average change from baseline through Week 2 (DAVG2) for HIV-1 RNA (log10 copies/mL) | Baseline to Week 2
  DAVG2 was defined as the time-weighted average between baseline value through the last available value up to week 2 minus the baseline value.

SECONDARY OUTCOMES:
Change from baseline in HIV-1 RNA (log10 copies/mL) | Baseline to Week 2
Change from baseline in CD4 cell count (cells/mm3) | Baseline to Week 2

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford Positive Care Program, Palo Alto, California
  - Protocare Trials Chicago Center for Clinical Trials, Chicago, Illinois
  - Rockefeller University Hospital, New York, New York